CLINICAL TRIAL: NCT06779409
Title: Comparing the Effects of Post Activation Potentiation on Vertical Jump Using High-Intensity Back Squat vs. Wingate Bike Test in Healthy Adults
Brief Title: Impact of the Wingate Test on Post-activation Potentiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00002860
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-03

CONDITIONS: Performance Enhancement; Muscle Activation
Keywords: post-activation potentiation; back squat; Wingate test; vertical jump; power; sport performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Back squat (Active Comparator): Participants will perform 2 sets of 3 repetitions at 85% of their 1 repetition maximum weight for the back squat
  Interventions: Other: Back squat
- Wingate test (Experimental): Participants will perform the Wingate bike test, with resistance at 7.5% of body weight, with a maximal effort for 30 seconds.
  Interventions: Other: Wingate test

INTERVENTIONS:
Other: Back squat — 2 sets of 3 repetitions of a back squat, set to 85% of the 1 repetition maximum weight
  Arms: Back squat
Other: Wingate test — 30 second maximal effort cycling test, with resistance at 7.5% bodyweight
  Arms: Wingate test

SUMMARY:
The goal of this trial is to see if using a maximal effort, short cycling test is better at activating muscles to improve vertical jump height compared to a maximal effort back squat. The study looks to answer three questions:

1. will the Wingate bike test create a different change in counter movement jump height compared to a back squat?
2. What is the best recovery period after each test where the counter movement jump is the highest?
3. What person-specific factors predict success of the Wingate bike test as a activation activity for the counter movement jump? Participants will visit the lab 3 times, once to give informed consent and measure their 1 repetition max (RM) back squat, and twice to perform each intervention and measure vertical jump height.

DETAILED DESCRIPTION:
Participants will be asked to come to the lab for three visits. On the first visit, they will perform informed consent, have anthropometrics taken, and will provide data to assess weightlifting history and factors that may influence the impact of each intervention. They will perform a 1 repetition max (RM) test for the back squat in order to properly dose the back squat potentiation activity. Visits 2 and 3 will be randomized; one will use the back squat (control) and the other will use the Wingate bike test (experimental) to potentiate vertical jump height as measured by the counter movement jump (CMJ). In each session, a warm up will be performed and the baseline CMJ will be performed. The intervention will be performed, either the 30 second Wingate protocol which is a maximal effort cycling test, or the back squat at a high percent of the 1 RM. The CMJ will be reassessed at 3, 6, and 9 minutes after completed each intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult
* successful completion of the physical activity readiness questionnaire plus
* at least 1 year of back squat weight training experience

Exclusion Criteria:

* inability to back squat at least 1.4 times body weight
* females with known pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Height | Visit 2 (1 week post- enrollment); visit 3 (2 weeks post-enrollment)
  Measured with the Counter Movement Jump (CMJ). This measures the vertical distance a participant is able to jump from a standing, stationary position. Video capture and motion analysis software will be used to analyze the jump and determine vertical displacement of a marker placed at the participants sacrum. Vertical jump height will be measured in meters.

SECONDARY OUTCOMES:
Years of resistance training experience | Collected at visit 1, upon enrollment into the study
  This factor will be collected to examine its predictive impact on the Wingate test's potentiation effect. The number of years of resistance training each participants has participated in will be collected.
One-Repetition Maximum Back Squat Strength | Collected at visit 1, upon enrollment into the study
  This factor will be collected to examine its predictive impact on the Wingate test's potentiation effect. The 1 repetition maximum weight in kilograms for the back squat exercise will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, DPT, Principal Investigator — Louisiana State University Health Sciences Center Shreveport
Locations (1):
- LSU Health Shreveport School of Allied Health Professions, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Available 3 months following publication of findings, no end date (link to be provided)
Access Criteria: Researchers wishing to access the data

REFERENCES:
- [Background] Sirieiro P, Nasser I, Dobbs WC, Willardson JM, Miranda H. The Effect of Set Configuration and Load on Post-Activation Potentiation on Vertical Jump in Athletes. Int J Exerc Sci. 2021 Aug 1;14(4):902-911. doi: 10.70252/CCLW6758. eCollection 2021. PMID 34567370
- [Background] Jo E, Judelson DA, Brown LE, Coburn JW, Dabbs NC. Influence of recovery duration after a potentiating stimulus on muscular power in recreationally trained individuals. J Strength Cond Res. 2010 Feb;24(2):343-7. doi: 10.1519/JSC.0b013e3181cc22a4. PMID 20072066
- [Background] Esformes JI, Bampouras TM. Effect of back squat depth on lower-body postactivation potentiation. J Strength Cond Res. 2013 Nov;27(11):2997-3000. doi: 10.1519/JSC.0b013e31828d4465. PMID 23442291
- [Background] Lowery RP, Duncan NM, Loenneke JP, Sikorski EM, Naimo MA, Brown LE, Wilson FG, Wilson JM. The effects of potentiating stimuli intensity under varying rest periods on vertical jump performance and power. J Strength Cond Res. 2012 Dec;26(12):3320-5. doi: 10.1519/JSC.0b013e318270fc56. PMID 23007485
- [Background] McCann MR, Flanagan SP. The effects of exercise selection and rest interval on postactivation potentiation of vertical jump performance. J Strength Cond Res. 2010 May;24(5):1285-91. doi: 10.1519/JSC.0b013e3181d6867c. PMID 20393352